CLINICAL TRIAL: NCT05679440
Title: Pulmonary Imaging-based Postural Ventilation in Patients With Severe COVID-19 - a Prospective, Non-randomized Controlled Study
Brief Title: Postural Changes and Severe COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wang xiaorong, Internal medicine physician, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RICU20230103
Record Dates: First submitted 2023-01-08; First posted 2023-01-11 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: COVID-19; pulmonary imaging; prone position; lateral position; prognosis
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: In the intervention group, arterial blood gases, heart rate, blood pressure, finger pulse oxygen saturation and inhaled oxygen concentration were collected 30 minutes before ventilation in different positions according to pulmonary imaging data (Time 1). Patients are ventilated in prone position (for patients with bilateral lung lesions), left/right lateral position, semi-prone position (for patients with unilateral lung lesions or those who cannot tolerate prone ventilation, so that the diseased lung is above and the healthy lung is below), supine position (for patients who cannot tolerate prone ventilation or lateral ventilation, etc.) according to the pulmonary imaging data. Arterial blood gases, heart rate, blood pressure, finger pulse oxygen saturation, and inhaled oxygen concentration were collected again when the patient was ventilated in the different positions for 2 hours (Time 2).
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients in the control group are ventilated in a comfortable position according to the principles of treatment and their wishes
- Intervention group (Experimental): Patients are ventilated in prone position (for patients with bilateral lung lesions), left/right lateral position, semi-prone position (for patients with unilateral lung lesions or those who cannot tolerate prone ventilation, so that the diseased lung is above and the healthy lung is below), supine position (for patients who cannot tolerate prone ventilation or lateral ventilation, etc.) according to the pulmonary imaging data.
  Interventions: Behavioral: Postural interventions based on pulmonary imaging

INTERVENTIONS:
Behavioral: Postural interventions based on pulmonary imaging — The main difference between the intervention group and the control group was the position during oxygen therapy. Patients in the intervention group were placed in the appropriate position for oxygen therapy according to pulmonary imaging, while patients in the control group were placed in the appropriate position for oxygen therapy according to conventional treatment principles and the patient's wishes.
  Arms: Intervention group

SUMMARY:
COVID-19 remains a widespread global epidemic, increasing morbidity, mortality, healthcare resource consumption, and socio-economic burden on patients worldwide. The onset of COVID-19 ranges from mild, self-limiting respiratory disease to severe progressive pneumonia, mainly acute respiratory distress syndrome (ARDS), with critically ill patients requiring admission to the intensive care unit (ICU).

Prone positioning has been shown to improve oxygenation and reduce complications and mortality in patients with severe ARDS. Prone position increases functional residual volume and chest wall elasticity, reduces dorsal segment edema in both lower lungs, facilitates uniform ventilation distribution, improves V/Q ratio, reduces alveolar shunts, and aids secretion drainage. In clinical practice, the prone position is mainly used for patients with diffuse bilateral lung lesions. However, it is less effective in unilateral or predominantly upper lung patients. Moreover, some patients are unable to tolerate prone ventilation. Therefore, we construct an individualized approach to postural oxygen therapy by guiding the patient's position based on the pulmonary imaging information.

A study on the optimal ventilation position for patients with severe COVID-19 will be conducted at the Department of Respiratory and Critical Care Medicine, Wuhan Union Hospital. The investigators enrolled adult patients (without endotracheal intubation) diagnosed with severe COVID-19 requiring oxygen therapy from 2023.01.10 to 2024.01.10. Patients were grouped into control and intervention groups according to current treatment protocol and pulmonary imaging combined with patients' wishes and degree of postural tolerance. Patients in the intervention group were ventilated in different positions according to pulmonary imaging, including prone, left/right lateral, supine, semi-recumbent, and seated. In contrast, patients in the control group were ventilated comfortably according to the treatment principles and their wishes. The primary observation was 28-day mortality. Secondary observations were oxygenation index (PaO2/FiO2) before and after a position change, endotracheal intubation rate, duration of respiratory support, length of hospital stay, and comfort in position.

DETAILED DESCRIPTION:
Study population:

Adult patients with severe COVID-19 requiring oxygen therapy who were not endotracheally intubated at the Department of Respiratory and Critical Care Medicine, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology were selected.

Diagnostic Criteria:

Diagnostic criteria for severe COVID-19: A diagnosis of severe COVID-19 is made when any of the following criteria are met.

1. Presence of shortness of breath with an RR ≥ 30 beats/min.
2. Finger oxygen saturation ≤93% on air inhalation at rest.
3. Oxygenation index (arterial partial pressure of oxygen/oxygen concentration) ≤ 300 mmHg (1 mmHg = 0.133 kPa), or arterial partial pressure of oxygen ≤ 60 mmHg when breathing air at rest.
4. Progressive worsening of clinical symptoms and pulmonary imaging showing the significant progression of >50% of the lesion within 24 to 48 hours.

Inclusion criteria:

(1)age ≥ 18 years; (2) admitted with a confirmed diagnosis of severe COVID-19; (3) Patients without endotracheal intubation requiring high flow nasal cannula, non-invasive ventilator, mask, nasal cannula assisted ventilation; (4) signed informed consent.

Exclusion criteria:

(1)hemodynamic instability; (2) unstable spinal fractures; (3) unstable pelvic or long bone fractures; (4) open abdominal wounds; (5) late pregnancy; (6) increased intracranial pressure due to a lesion in the head and neck that obstructs cerebral venous drainage.

Content and methods:

Patients who met the study criteria were selected according to the inclusion and exclusion criteria. Adult patients with confirmed severe COVID-19 and requiring oxygen therapy were admitted to the Department of Respiratory and Critical Care Medicine, Wuhan Union Hospital, from 2023.01.10 to 2024.01.10 without tracheal intubation were included. Informed consent was obtained from the patients and their families and signed. Investigators collected baseline data on demographics, anthropometrics, concomitant diseases, arterial blood gases on admission, and oxygen therapy modalities and parameters for all patients. After inclusion in the study, all patients were grouped into control and intervention groups according to the treatment protocol and pulmonary imaging in combination with the patient's wishes and tolerance of the position. According to pulmonary imaging data, in the intervention group, arterial blood gases, heart rate, blood pressure, finger pulse oxygen saturation, and inhaled oxygen concentration were collected 30 minutes before ventilation in different positions (Time 1). Patients are ventilated in a prone position (for patients with bilateral lung lesions), left/right lateral position, semi-prone position (for patients with unilateral lung lesions or those who cannot tolerate prone ventilation, so that the diseased lung is above and the healthy lung is below), supine position (for patients who cannot tolerate prone ventilation or lateral ventilation, etc.) according to the pulmonary imaging data. Arterial blood gases, heart rate, blood pressure, finger pulse oxygen saturation, and inhaled oxygen concentration were collected again when the patient was ventilated in different positions for 2 hours (Time 2). Patients in the control group are ventilated comfortably according to the treatment principles and their wishes. All patients were homogenized regarding medication and ventilation during their hospitalization, except for the choice of position during ventilation. The primary observation was 28-day mortality. Secondary observations were oxygenation index (PaO2/FiO2) before and after a position change, tracheal intubation rate, duration of respiratory support, length of stay, and comfort in position.

The primary information recorded during the patient's hospitalization included: gender, age, concomitant diseases, history of smoking, alcohol consumption, body mass index (BMI), position and duration of ventilation. Prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (INR), B-type natriuretic peptide (BNP), D dimer, leukocytes, platelets, lymphocytes, C-reactive protein (CRP), procalcitonin (PCT), ferritin, inflammatory factors, liver function, renal function; imaging information including lung CT; and disease-related scores, including acute physiology and chronic health inquiry (APACHE) Ⅱ score, Glasgow Coma Scale (GCS), sequential organ failure assessment (SOFA) score, etc.

Choice of ventilation modality:

All patients included in this study were non-endotracheally intubated patients with severe COVID-19 who were routinely administered oxygen therapy during hospitalization. Depending on the patient's condition, the oxygen therapy modalities used during the study included the high-flow nasal cannula (HFNC), non-invasive ventilator, face mask, and nasal cannula. Patients were ventilated by the same method before and after changing positions.

Clinical Outcomes:

Primary clinical outcome: 28-day mortality. Secondary clinical outcomes: oxygenation index (PaO2/FiO2) before and after a position change, endotracheal intubation rate, duration of respiratory support, length of stay, hospital costs, and comfort in position.

Sample size:

The sample size for this project was calculated using the chi-square Contingency Table (Chi-Square Tests) for the two rates in PASS 15.0 software. A literature review revealed that the current use of prone ventilation in patients with severe COVID-19 is 67.36%. In the study, the test level was α=0.05, and the test efficacy was 1 - β=0.9. The final sample size was 100 cases, considering that some patients dropped out in the middle of the study or could not tolerate it.

Statistical analysis and statistical methods:

The data obtained during the study were pre-collated. For continuous data, normality tests were first performed. If all groups met normality, the Student's t-test was used for comparison between groups. Otherwise, the non-parametric Wilcoxon rank sum test was considered. For categorical variables, the χ2 test was used. Statistically significant data were subjected to multivariate logistic regression analysis. Receiver operating characteristic (ROC) and Delong's method were used to analyze the effect of oxygen therapy in different positions on the prognosis of patients with severe COVID-19, with a difference considered statistically significant at P < 0.05.

Statistical analysis of all data was performed through SPSS (IBM SPSS Statistics 26.0, SPSS Inc., Chicago, IL) and R language (version 4.1.3, www.R-project.org/). All statistical tests were two-sided, and statistical significance was set at 0.05.

Safety evaluation:

This study investigates the effect on oxygen saturation and prognosis of patients with severe COVID-19 when oxygen therapy is administered in prone, lateral, supine, and semi-recumbent positions. Healthcare staff also make rounds during the change of position and will promptly deal with any dislodgement of the line to minimize harm to the patient and not cause additional harm to the patient. In summary, this study was safe in its implementation.

Adverse events:

In the event of the patient's condition deterioration or respiratory distress during the program, treatment will be adjusted according to the patient's condition. Investigators will monitor the patient's condition in real-time and perform endotracheal intubation if necessary to minimize harm to the patient. The decision to withdraw from this clinical study will be based on the patient's family's wishes.

Informed Consent Process:

Informed consent is completed before the subject's participation and continues throughout the study. The ethics committee agrees to inform consent, and the subject reads the informed consent form. The investigator will explain the process, answer questions from the subject, and inform the subject of the possible risks and their rights. Before agreeing to participate, the subject may discuss this with a family member or guardian. The researcher must inform the subject that participation in the study is voluntary and that they may withdraw from the study at any time during the study. A copy of the informed consent form may be provided to the research subject for retention. The rights and welfare of the research subjects will be protected, and it is stressed that the quality of their medical care will not be compromised by their refusal to participate in the study.

Privacy Protection:

All information collected in this study is managed with particular confidentiality, and any study information cannot be disclosed to unauthorized third parties without prior approved consent.

Quality control and quality assurance:

All clinical data in this project were obtained from the inpatient case management system of Union Hospital, Tongji Medical College, Huazhong University of Science and Technology. Patients with COVID-19 were screened according to the inclusion criteria, and clinical data were collected. The data collected did not include the content of the patient's privacy section, and all quality management and quality control were supervised and managed by one person. The investigators received systematic methodological training at the start of the project.

Data collection and management:

The data for this study were obtained from the medical records of inpatients within the Wuhan Union Hospital. All data were transparent, accurate, and traceable. A clinical database was established during the study, which was password-protected and complied with logical proofreading procedures.

Study data retention:

All raw data and original documentation required for this project will be retained until at least three years after the end of the clinical trial, and permission should be obtained before destruction.

Declarations of interest:

The investigators have disclosed that they do not have any conflicts of interest.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admitted with a confirmed diagnosis of COVID-19 severe pneumonia
* Patients without endotracheal intubation requiring high flow nasal cannula, non-invasive ventilator, mask, nasal cannula assisted ventilation
* Signed informed consent

Exclusion Criteria:

* Hemodynamic instability
* Unstable spinal fractures
* Unstable pelvic or long bone fractures
* Open abdominal wounds
* Late pregnancy
* Increased intracranial pressure due to a lesion in the head and neck that obstructs cerebral venous drainage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-01-10 (Estimated); Study Completion 2024-01-10 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | 28 days
  Comparison of patients' deaths 28 days after admission.

SECONDARY OUTCOMES:
Endotracheal intubation rate | From the date of the non-randomised cohort study until the date of death or discharge from hospital for any reason, whichever comes first, with a maximum assessment period of 3 months
  Patients require endotracheal intubation and mechanical ventilation due to deterioration or exacerbation of their condition during hospitalisation.
Length of respiratory support | From the date of the non-randomised cohort study until the date of death or discharge from hospital for any reason, whichever comes first, with a maximum assessment period of 3 months
  Time spent by patients in hospital on oxygen therapy using high-flow nasal cannulae, non-invasive ventilators, face masks and nasal cannulae.
Length of hospital stay | From the date of the non-randomised cohort study until the date of death or discharge from hospital for any reason, whichever comes first, with a maximum assessment period of 3 months
  Length of time patients are treated in hospital.
Hospital costs | From the date of the non-randomised cohort study until the date of death or discharge from hospital for any reason, whichever comes first, with a maximum assessment period of 3 months
  Costs incurred during the patient's stay in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Wang, Ph.D., M.D., Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
In this study, we will share parts of the study design such as Study Protocol, Statistical Analysis Plan (SAP) and Informed Consent Form (ICF).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We will share the data 6 months after the end of the study, which lasts for 6 months.
Access Criteria: Data were obtained through the Principal Investigator of this study upon reasonable request.

REFERENCES:
- [Background] Tu GW, Liao YX, Li QY, Dong H, Yang LY, Zhang XY, Fu SZ, Wang RL. Prone positioning in high-flow nasal cannula for COVID-19 patients with severe hypoxemia: a pilot study. Ann Transl Med. 2020 May;8(9):598. doi: 10.21037/atm-20-3005. No abstract available. PMID 32566624
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Liang WH, Guan WJ, Li CC, Li YM, Liang HR, Zhao Y, Liu XQ, Sang L, Chen RC, Tang CL, Wang T, Wang W, He QH, Chen ZS, Wong SS, Zanin M, Liu J, Xu X, Huang J, Li JF, Ou LM, Cheng B, Xiong S, Xie ZH, Ni ZY, Hu Y, Liu L, Shan H, Lei CL, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Cheng LL, Ye F, Li SY, Zheng JP, Zhang NF, Zhong NS, He JX. Clinical characteristics and outcomes of hospitalised patients with COVID-19 treated in Hubei (epicentre) and outside Hubei (non-epicentre): a nationwide analysis of China. Eur Respir J. 2020 Jun 4;55(6):2000562. doi: 10.1183/13993003.00562-2020. Print 2020 Jun. PMID 32269086
- [Background] Grasselli G, Zangrillo A, Zanella A, Antonelli M, Cabrini L, Castelli A, Cereda D, Coluccello A, Foti G, Fumagalli R, Iotti G, Latronico N, Lorini L, Merler S, Natalini G, Piatti A, Ranieri MV, Scandroglio AM, Storti E, Cecconi M, Pesenti A; COVID-19 Lombardy ICU Network. Baseline Characteristics and Outcomes of 1591 Patients Infected With SARS-CoV-2 Admitted to ICUs of the Lombardy Region, Italy. JAMA. 2020 Apr 28;323(16):1574-1581. doi: 10.1001/jama.2020.5394. PMID 32250385
- [Background] Munshi L, Del Sorbo L, Adhikari NKJ, Hodgson CL, Wunsch H, Meade MO, Uleryk E, Mancebo J, Pesenti A, Ranieri VM, Fan E. Prone Position for Acute Respiratory Distress Syndrome. A Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2017 Oct;14(Supplement_4):S280-S288. doi: 10.1513/AnnalsATS.201704-343OT. PMID 29068269
- [Background] Guerin C, Beuret P, Constantin JM, Bellani G, Garcia-Olivares P, Roca O, Meertens JH, Maia PA, Becher T, Peterson J, Larsson A, Gurjar M, Hajjej Z, Kovari F, Assiri AH, Mainas E, Hasan MS, Morocho-Tutillo DR, Baboi L, Chretien JM, Francois G, Ayzac L, Chen L, Brochard L, Mercat A; investigators of the APRONET Study Group, the REVA Network, the Reseau recherche de la Societe Francaise d'Anesthesie-Reanimation (SFAR-recherche) and the ESICM Trials Group. A prospective international observational prevalence study on prone positioning of ARDS patients: the APRONET (ARDS Prone Position Network) study. Intensive Care Med. 2018 Jan;44(1):22-37. doi: 10.1007/s00134-017-4996-5. Epub 2017 Dec 7. PMID 29218379
- [Background] Gattinoni L, Taccone P, Carlesso E, Marini JJ. Prone position in acute respiratory distress syndrome. Rationale, indications, and limits. Am J Respir Crit Care Med. 2013 Dec 1;188(11):1286-93. doi: 10.1164/rccm.201308-1532CI. PMID 24134414
- [Background] Hewitt N, Bucknall T, Faraone NM. Lateral positioning for critically ill adult patients. Cochrane Database Syst Rev. 2016 May 12;2016(5):CD007205. doi: 10.1002/14651858.CD007205.pub2. PMID 27169365
- [Background] Le MQ, Rosales R, Shapiro LT, Huang LY. The Down Side of Prone Positioning: The Case of a Coronavirus 2019 Survivor. Am J Phys Med Rehabil. 2020 Oct;99(10):870-872. doi: 10.1097/PHM.0000000000001530. PMID 32657818
- [Background] Pan C, Chen L, Lu C, Zhang W, Xia JA, Sklar MC, Du B, Brochard L, Qiu H. Lung Recruitability in COVID-19-associated Acute Respiratory Distress Syndrome: A Single-Center Observational Study. Am J Respir Crit Care Med. 2020 May 15;201(10):1294-1297. doi: 10.1164/rccm.202003-0527LE. No abstract available. PMID 32200645